CLINICAL TRIAL: NCT01883622
Title: Glucose Fluctuations During Gestation: an Additional Tool for a Better Monitoring of Pregnancy Complicated by Diabetes
Brief Title: Glucose Variability in Pregnancy Complicated by Diabetes
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: GES03
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Gestational Diabetes; Continuous Glucose Monitoring; Glycemic Variability
Keywords: diabetes; pregnancy; glucose variability; continuous glucose monitoring (CGM); gestational diabetes mellitus (GDM)
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Type 1 diabetes: Pregnant women affected by type 1 diabetes mellitus
- GDM: Pregnant women affected by gestational diabetes mellitus
- Healthy: Healthy pregnant women

SUMMARY:
Continuous glucose monitoring (CGM) methods provide details of magnitude and duration of glucose fluctuations, giving a unique insight on daily blood sugar control. Limited data are available on glucose variability (GV) in pregnancy. The aim of this study was to assess GV in normal pregnant women and cases of type 1 diabetes mellitus or gestational diabetes (GDM), and its possible association with HbA1c.

DETAILED DESCRIPTION:
Recent evidence in the literature suggests that glucose variability, characterized by extreme glucose excursions, may overlap with HbA1c levels in determining the risk of diabetes-related complications. Fluctuating blood glucose levels prompt an increase in free radicals and endothelial dysfunction, which are the links between hyperglycemia and the activation of pathological pathways that lead to tissue damage. Reece and Homko postulated an association between maternal hyperglycemia-induced oxygen free radical overproduction and fetal abnormalities, with the onset of diabetes-related embryopathy.Numerous studies have demonstrated that macrosomia and congenital malformations relate to glycemic control. In one study, 48-hour continuous glucose monitoring (CGM) of diurnal glucose profiles in pregnant women with type 1 diabetes was more sensitive than HbA1c alone in identifying an increased risk of offspring with congenital malformations. Such studies give the impression that transient hyperglycemic spikes in pregnant patients with diabetes can cause a high incidence of fetal overweight, regardless of whether or not the mother has chronic hyperglycemia. Glucose variability is still a factor that has been inadequately studied in pregnancies complicated by diabetes, and little is known about its relationship with maternal-fetal outcomes.A number of studies have demonstrated the utility of CGM for monitoring diabetes in pregnancy , but none have focused the attention on the importance of glucose fluctuations during gestation. Meanwhile, there has been a rapid increase in the number of new glucose variability indicators considered, although none of them seems to be definitively reliable.

A better understanding of the pattern of blood glucose fluctuations in all the three trimesters of pregnancy, could help us to optimize glycemic control in pregnant women with diabetes.

The aim of this study was therefore to assess glucose variability throughout the three trimesters of pregnancy in healthy women and in cases of type 1 diabetes mellitus or gestational diabetes, identifying the more representative and useful indicators of glucose fluctuations, to provide more accurate clinical informations along with HbA1c and beyond.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 1 diabetes or GDM
* able to become familiar with glucose monitoring methodologies

Exclusion Criteria:

* type 2 diabetes
* pre-gestational BMI > 35 Kg/m2
* HbA1c > 8% for type 1 diabetic pregnant women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Outpatient pregnant women enrolled at three Italian diabetes clinics (Padua, Pisa and Florence)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2004-01; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Glucose variability indexes during first, second and third trimester of pregnancy | 9 months
  Patients wore underwent continuous glucose monitoring for 2 days in each trimester of pregnancy. As indexes of glucose variability we considered: the mean amplitude of glucose excursion (MAGE); the total standard deviation (SD); the interquartile range (IQR); the continuous overlapping net glycemic action (CONGA1), calculated at 1 hour. The low blood glucose index (LBGI) and high blood glucose index (HBGI) were also calculated.

SECONDARY OUTCOMES:
Association between HbA1c and glucose variability indicators in the three trimesters pf pregnancy, in the three groups of women | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Annunziata Lapolla, MD, Study Chair — Department of Medicine, University of Padova
Locations (3):
- Italy (3):
  - Department of Gynecology, Perinatology and Human Reproduction, University of Florence, Florence
  - Department of Medicine, University of Padua, Padua
  - Department of Endocrinology and Metabolic Diseases, University of Pisa, Pisa

REFERENCES:
- [Background] Dalfra MG, Sartore G, Di Cianni G, Mello G, Lencioni C, Ottanelli S, Sposato J, Valgimigli F, Scuffi C, Scalese M, Lapolla A. Glucose variability in diabetic pregnancy. Diabetes Technol Ther. 2011 Aug;13(8):853-9. doi: 10.1089/dia.2010.0145. PMID 21751862
- [Background] Kerssen A, de Valk HW, Visser GH. Forty-eight-hour first-trimester glucose profiles in women with type 1 diabetes mellitus: a report of three cases of congenital malformation. Prenat Diagn. 2006 Feb;26(2):123-7. doi: 10.1002/pd.1340. PMID 16463292
- [Background] Di Cianni G, Miccoli R, Volpe L, Lencioni C, Del Prato S. Intermediate metabolism in normal pregnancy and in gestational diabetes. Diabetes Metab Res Rev. 2003 Jul-Aug;19(4):259-70. doi: 10.1002/dmrr.390. PMID 12879403